CLINICAL TRIAL: NCT01065168
Title: Serial Measurement of Serum Antimullerian Hormone in Women Undergoing Laparoscopic Cystectomy of Endometrioma
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Singpetch Suksompong, Mahidol University
Other Study IDs: si637/2008
Record Dates: First submitted 2010-02-06; First posted 2010-02-09 (Estimated); Last update posted 2010-02-17 (Estimated); Status verified 2009-01

CONDITIONS: Endometriosis
Keywords: endometriosis; endometrioma; antimullerian hormone; cystectomy
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- endometrioma: ovarian endometrioma undergoing cystectomy

SUMMARY:
The purpose of this trial is to study ovarian reserve after laparoscopic endometrioma cystectomy by measuring antimullerian hormone. The measurements were measured before the surgery and one week and three months after the surgery.

DETAILED DESCRIPTION:
Antimullerian hormone will be obtained in patients with ovarian endometrioma before laparoscopic cystectomy is done. The measurements were compared with antimullerian hormone after one week and three months after the surgery. Forty three patients will be included in this study.

ELIGIBILITY:
Inclusion Criteria:

* 20-40 years
* ovarian endometrioma > or = 3 cms
* laparoscopic cystectomy treatment

Exclusion Criteria:

* previous ovarian surgery
* other ovarian pathology
* previous drugs or hormonal treatment for endometrioma

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: ovarian endometrioma performed laparoscopic cystectomy
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2009-01; Primary Completion 2010-01 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
Ovarian reserve before and after ovarian endometrioma cystectomy. | one week and three months

CONTACTS AND LOCATIONS:
Overall Officials: Singpetch Suksompong, Doctor, Principal Investigator — Mahidol University